CLINICAL TRIAL: NCT01025713
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Trial to Assess the Safety, Tolerability, and Pharmacokinetics of GS 9411 in Subjects With Cystic Fibrosis (CF)
Brief Title: A Phase 1 Trial to Assess the Safety, Tolerability, and Pharmacokinetics of GS 9411 in Subjects With Cystic Fibrosis (CF)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development program terminated.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-221-0106
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis; Mucociliary Clearance
Keywords: Cystic Fibrosis; CF; Mucociliary Clearance; Epithelial Sodium Channel Inhibitor; ENaC Inhibitor; Airway Hydration; Amiloride
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): GS-9411 2.4 mg
  Interventions: Drug: GS-9411
- 2 (Experimental): GS-9411 4.8 mg
  Interventions: Drug: GS-9411
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-9411 — Inhaled GS-9411
  Arms: 1; 2
Drug: Placebo — Inhaled Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of GS-9411 in patients with Cystic Fibrosis. GS-9411 is a sodium channel inhibitor, that may restore airway hydration and mucociliary clearance in the lung.

DETAILED DESCRIPTION:
GS-9411 is being evaluated as a potential therapy to improve airway hydration and mucociliary clearance in patients with cystic fibrosis. This study is evaluating the safety and tolerability of 2 dose levels of GS-9411 as an inhaled product, compared to a matched placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 65 years
* Patients with diagnosis of CF as confirmed by at least one of the following:
* Documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis test OR
* Documented sweat sodium test ≥ 60 mmol/L OR
* Abnormal nasal potential difference test OR
* At least one well-characterized disease-causing genetic mutation in the CF transmembrane conductance regulatory (CFTR) gene AND
* Accompanying symptoms characteristic of CF
* Normal (or abnormal but not clinically significant) electrocardiogram (ECG)
* Normal intraocular pressure (IOP) between 10 and 21 mm Hg at Screening.
* Normal (or abnormal but not clinically significant) blood pressure (BP) and heart rate (HR) in the absence of any medications for hypertension; these will be measured after the subject has rested supine for 3 minutes; normal BP is taken to be 90 to 140 mm Hg systolic and 50 to 89 mm Hg diastolic; normal HR is taken to be 40 to 100 beats per minute (bpm)
* Able to communicate well with the investigator and to comply with the requirements of the entire study
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form
* Nonsmokers for at least 180 days (6 months) prior to Screening
* Must be willing to abstain from alcohol and strenuous exercise during the 48 hours prior to Screening, 72 hours prior to initial dosing, and during the study
* Forced expiratory volume in 1 second (FEV1) ≥ 50% predicted normal for age, gender, and height at Screening as per Knudson et al
* Stable regimen of oral CF medications, dornase alfa, and physiotherapies for the period 28 days prior to Screening; those subjects taking continuous (non-cycling) inhaled antibiotics for prophylaxis must be on a stable regimen of these drugs for at least 90 days prior to Screening
* Subjects must be in the off-phase of any cyclical inhaled antibiotic treatment regimen
* Must test negative for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV) at Screening
* Male subjects who are sexually active must be willing to use effective barrier contraception (e.g., condom) during heterosexual intercourse from Day -1 through completion of the study and continuing for at least 90 days from date of last dose of study drug
* Male subjects must refrain from sperm donation from Day -1 through completion of the study and continuing for at least 90 days from the date of last dose of study drug
* Nonlactating females. Females on hormone replacement therapy (estrogen/progesterone) or contraceptive therapy must be stabilized on a product and dose for at least 90 days prior to Screening
* Females must have a negative serum gonadotropin pregnancy test at Screening and Day -1
* Nonpregnant females of childbearing potential must agree to use highly effective (<1% failure rate) contraception during heterosexual intercourse from Screening, throughout the study, and for at least 30 days following the last dose of study drug
* Glomerular filtration rate (GFR) of < 60 mL/min/1.73m2 at Screening (GFR to be calculated using the Cockcroft-Gault equation), and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3× upper limits of normal (ULN)
* Chest radiograph at Screening without significant acute findings (e.g., infiltrates [lobar or diffuse interstitial], pleural effusion, pneumothorax); or chest radiograph, CT, or MRI obtained within the 90 days prior to Screening without acute findings or significant intercurrent illness; chronic, stable findings (e.g., chronic scarring or atelectasis) are allowed. A chest radiograph obtained and interpreted between Screening and Day 1 is also acceptable for determining eligibility.

Exclusion Criteria:

* Administration of any investigational drug or device in the 28 days prior to Screening
* A need for any new medication during the period 28 days before first dosing with study drug, except those deemed by the principal investigator/clinical investigator not to interfere with the outcome of the study
* Subjects who routinely use inhaled hypertonic saline must discontinue use for at least 14 days prior to clinic admission and for the duration of the study
* Use of trimethoprim or high dose ibuprofen (> 800 mg/day) during the 28 days prior to first dosing
* Serious adverse reaction or hypersensitivity to any drug
* Existence of any surgical or medical condition which, in the judgment of the clinical investigator, might interfere with the absorption, distribution, metabolism, or excretion of the drug
* Lactating females
* History of airway intolerance to hypertonic saline
* History of lung transplantation
* History of a positive test for Burkholderia cepacia
* History of cirrhosis or ascites
* History of clinically significant adrenal disease
* History of congestive heart failure diagnosed clinically or with documented left ventricular ejection fraction (LVEF) ≤ 40%
* History of glaucoma
* Consumption of drugs and/or herbal preparations capable of inducing hepatic enzyme metabolism (e.g., barbiturates, rifampicin, carbamazepine, phenytoin, primidone, or St. John's Wort) within 28 days (or 5 half-lives of inducing agent, whichever is longer) of Screening
* Subjects requiring any of the following drugs in the 28 days prior to Screening: diuretics (e.g., spironolactone, amiloride, thiazide), ACE inhibitors, angiotensin receptor blockers, oral corticosteroids, or medicines for hypertension
* Donation or loss of greater than 400 mL of blood in the period 90 days (3 months) prior to Screening
* Major surgery within 180 days (6 months) of Screening
* Hemoglobin levels < 120 g/L in females or < 130 g/L in males taken at Screening and at Day -1
* Serum potassium > 5 mEq/L taken at Screening and at Day -1
* Poor venous access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of escalating doses of inhaled GS-9411 in subjects with CF. | 5 Days

SECONDARY OUTCOMES:
To assess the pharmacokinetics (PK) of GS-9411 and its metabolites, in plasma, urine, and sputum after single inhaled doses. | 5 Days

CONTACTS AND LOCATIONS:
Overall Officials: John Wilson, MD, Principal Investigator — The Alfred
Locations (1):
- Nucleus Network, Ltd., Melbourne, Victoria, Australia